CLINICAL TRIAL: NCT04285801
Title: Critically Ill Patients With COVID-19 in Hong Kong: a Multicentre Observational Cohort Study
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lowell Ling, Clinical Lecturer, Chinese University of Hong Kong
Other Study IDs: 2020.059
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 infection: critically ill patients with COVID-19 infection

SUMMARY:
The purpose of this case series is to describe the characteristics, organ dysfunction and support and 2 week outcomes of critically ill patients with nCov infection.

DETAILED DESCRIPTION:
The 2019 novel-coronavirus (2019-nCov) is the cause of a cluster of unexplained pneumonia that started in Hubei province in China 1. It has manifest into a global health crisis with escalating confirmed cases and spread across 15 countries. Whilst it is currently an epidemic in China, The World Health Organization (WHO) Global Level risk assessment is set at high 2.

Sequencing showed that 2019-nCov is similar to bat severe acute syndrome (SARS)-related coronaviruses found in Chinese horseshoe bats 3. This is compatible with the initial epidemiological link with a local wet market which sells bats. Furthermore, data sharing and sequencing data has facilitated development of accurate diagnostic tests.

In contrast, our current understanding of the epidemiological and clinical features of 2019-nCov is limited. In a case series of 41 hospitalized patients with confirmed infection, at least 30% of these patients required critical care admission. These patients developed severe respiratory failure and 10% required mechanical ventilation and 5% needed extracorporeal membrane oxygenation support. More worryingly 2019-nCov infection was associated with 15% mortality. Although these figures are likely overestimates due to unreported mild cases, there is currently no effective treatment. The optimal supportive care for patients with severe 2019-nCov infection is a research priority.

The spread of the 2019-nCov epidemic to Hong Kong has started. Patients have been admitted to the Intensive Care Unit for multiorgan dysfunction. Currently there are no published data focused specifically on critically ill patients with nCov infection. The purpose of this case series is to describe the characteristics, organ dysfunction and support and 2 week outcomes of critically ill patients with nCov infection.

ELIGIBILITY:
Inclusion Criteria:

* admission to ICU
* adult (≥18 years old)
* confirmed case of 2019-nCov infection by 2019-nCov RNA by reverse transcription polymerase chain reaction , isolation in cell culture of 2019-nCov from a clinical specimen or serum antibody to 2019-nCov

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All critically ill patients with confirmed COVID-19 infection in Hong Kong
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
28 day mortality | 28 days
  survival or death at 28 days

SECONDARY OUTCOMES:
vasopressor days | 28 days
  days on vasopressor
days on mechanical ventilation | 28 days
  days on mechanical ventilation during ICU stay
sequential organ function assessment score | daily for first 5 days
  daily sequential organ function assessment score (0 minimum to 24 maximum), higher scores worse organ function
ECMO use | 28 days
  Percentage of patients requiring ECMO during ICU stay.
percentage nitric oxide use | 28 days
  percentage of patients requiring nitric oxide during ICU stay.
percentage free from oxygen supplement | 28 days
  percentage not requiring oxygen therapy

CONTACTS AND LOCATIONS:
Locations (3):
- Hong Kong (3):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No